CLINICAL TRIAL: NCT03652701
Title: Hair Up Prospective Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: sponsor discretion
Sponsor: Shmuel Gonen Technologies Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLPR-001-0002
Record Dates: First submitted 2018-06-27; First posted 2018-08-29 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Hair Loss
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hair Up (Experimental)
  Interventions: Other: Hair Up
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Hair Up — Herbal topical
  Arms: Hair Up
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The objective of this study is to assess the performance of Hair Up on female pattern hair shedding and regrowth. 58 adult female patients suffering from hair loss will be evaluated in a single center prospective study

ELIGIBILITY:
Inclusion Criteria:

* Women who report hair loss during the past 3 months prior to the study

Exclusion Criteria:

* Disorders and medications affecting hair loss/growth, pregnancy, scarring alopecia

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of hair loss | 1 month
  Pull test

SECONDARY OUTCOMES:
Assessment of hair regrowth | 3 months
  Photographic evaluation of the change in hair density according to the Savin score (scale of 1-mild to 9-severe)
Quality of life questionnaire | 3 months
  Assessment of quality of life byThe Women's Androgenetic Alopecia Quality of Life Questionnaire (WAAQOL)

IPD SHARING:
Plan to Share IPD: Undecided